CLINICAL TRIAL: NCT02609763
Title: Live Validation of the Lower Eyelid Steatoblepharon Severity (LESS) Scale
Status: Completed | Type: Observational
Sponsor: Topokine Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TPK-SCALE-03
Record Dates: First submitted 2015-11-16; First posted 2015-11-20 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Steatoblepharon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This observational study will test the inter-rater and test-retest reliability of the LESS scale in a live context.

ELIGIBILITY:
Inclusion Criteria:

* Must provide informed consent

Exclusion Criteria:

* Unable or unwilling to complete study procedures

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible adults with varying degrees of lower eyelid steatoblepharon
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
LESS score (Clinician-Reported) | Eyelids will be assessed on one day only (cross-sectional study)